CLINICAL TRIAL: NCT04536688
Title: A Phase 1b, Multicenter, Open-Label, Adaptive Design Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RGLS4326 Administered Via SC Injection to Patients With Autosomal Dominant Polycystic Kidney Disease
Brief Title: A Study of RGLS4326 in Patients With Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regulus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RGLS4326-03
Record Dates: First submitted 2020-08-24; First posted 2020-09-03 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Polycystic Kidney Disease, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Intervention Model Description: Cohorts will be enrolled and treated sequentially. Dosing decisions will be made based on prior cohort's safety and biomarker data. Six to 9 subjects will be enrolled in each cohort based on the magnitude and/or variability of the increase in PC1 and PC2 or to allow for replacement of subjects that do not complete the study. The highest dose (1 mg/kg) will be administered in cohort 1. If the Sponsor determines that the increase in PC1 and PC2 from baseline for cohort 1 is inadequate, the study may be stopped for futility. If the Sponsor determines that the increase from baseline for cohort 1 is adequate, then 0.3 mg/kg will be administered in cohort 2. Based on the increase of PC1 and PC2 from baseline in cohort 2, Sponsor may determine a higher dose needs to be evaluated, then 0.5 mg/kg will be administered in cohort 3. If the Sponsor determines that lower dose needs to be evaluated, then 0.1 mg/kg will be administered in cohort 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RGLS4326 1 mg/kg Q2W (Experimental): Eligible participants will receive subcutaneous injection of 1 mg/kg of RGLS4326 every other week for 4 doses
  Interventions: Drug: RGLS4326
- RGLS4326 0.3 mg/kg Q2W (Experimental): Eligible participants will receive subcutaneous injection of 0.3 mg/kg of RGLS4326 every other week for 4 doses
  Interventions: Drug: RGLS4326
- RGLS4326 0.1 or 0.5 mg/kg Q2W (Experimental): Eligible participants will receive subcutaneous injection of 0.1 or 0.5 mg/kg of RGLS4326 every other week for 4 doses
  Interventions: Drug: RGLS4326

INTERVENTIONS:
Drug: RGLS4326 — Solution for subcutaneous injection

SUMMARY:
Primary Objective

• To assess the dose response relationship between RGLS4326 and ADPKD biomarkers

Secondary Objectives

* To characterize the pharmacokinetic (PK) properties of RGLS4326 in plasma and urine
* To assess the safety and tolerability of RGLS4326

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, adaptive design dose-ranging study to evaluate ADPKD biomarkers, PK, safety, tolerability, and pharmacodynamics (PD) of RGLS4326 administered via SC injection to patients with ADPKD. The goal is to assess the dose response relationship between RGLS4326 and ADPKD biomarkers. The study will consist of three sequential cohorts with approximately 18 to 27 subjects total.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ADPKD patients 18 to 70 years old
* Class 1C, 1D, or 1E Mayo Imaging Classification of ADPKD (based upon prior MRI or CT Scan or MRI obtained during screening)
* Estimated GFR at Screening between 30 to 90 mL/min/1.73 m^2 calculated by the investigator using the Chronic Kidney Disease Epidemiology Collaboration equation (CKD-EPI)
* Body mass index (BMI) between 18 and 35 kg/m^2
* If the patient has hypertension, the antihypertensive regimen must be stable for at least 28 days prior to randomization and the blood pressure adequately controlled prior to randomization
* Female patients of childbearing potential must not be lactating and must have no plans to become pregnant during the course of the study through 28 days after the last dose of study drug. Female patients of childbearing potential who are heterosexual must agree to use one of the following methods of contraception considered to be highly effective (i.e., results in <1% failure rate when used consistently and correctly) from screening through 28 days after the last dose of study drug:

  * Intrauterine device (IUD) or intrauterine system (IUS) in place for at least 3 months prior to first dose
  * Partner has had a vasectomy. Vasectomy in the partner is only considered to be highly effective provided the partner is the sole sexual partner of the female patient of childbearing potential and the vasectomized partner has had a medical assessment of the surgical success.
  * Stable hormonal contraception associated with inhibition of ovulation (with approved oral, transdermal, or depot regimen) for at least 3 months prior to first dose
  * Bilateral tubal occlusion
* Female patient of non-childbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to the first dose of study drug:

  * Hysterectomy
  * Bilateral oophorectomy
  * Bilateral tubal occlusion
  * Bilateral salpingectomy or be postmenopausal with no periods for at least 1 year prior to the first dose of study drug.
* Male patients must agree to use a condom during heterosexual intercourse and to not have unprotected sexual intercourse with a female who is pregnant or breastfeeding from screening through 28 days after the last dose of study drug; and must agree to refrain from sperm donation for at least 90 days after the last dose of study drug
* Screening hematology and clinical chemistries must meet the following criteria:

  * Platelets >150 x 10^9/L
  * Total white blood cell (WBC) count >3.0 x 10^9/L and absolute neutrophil count >1.5 x 10^9/L
  * Hemoglobin >12 g/dL for females and >13.5 g/dL for males
  * Total and direct bilirubin <1.5x upper limit of normal (ULN), unless elevated bilirubin is associated with a known benign condition (e.g., Gilbert's syndrome)
  * Alanine aminotransferase (ALT) <1.5x ULN
  * Aspartate aminotransferase (AST) <1.5x ULN
  * Alkaline phosphatase (ALP) <1.5x ULN
  * Gamma-glutamyl transferase (GGT) <2x ULN Note: At the discretion of the Investigator, screening laboratory testing may be repeated once to confirm out of range (exclusionary) results.
* Able to understand all study procedures in the informed consent form (ICF) and willing to comply with all aspects of the protocol

Exclusion Criteria:

* Administration of tolvaptan in the 28 days before randomization
* Participation in another investigational interventional study within 28 days or 5 half-lives, whichever is longer, before randomization (e.g., bardoxolone, lixivaptan, tesevatinib, venglustat)
* A history of drug and/or alcohol abuse within the past year
* Active infection of the urinary tract (e.g., kidney, bladder, etc.)
* Known hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Only one kidney or kidney transplant recipient.
* Patient has concurrent medical condition (e.g., significant infection, other kidney disease, neurologic condition such as seizures, etc.) or social situation that may either present a safety risk or noncompliance with the study procedures
* History of active malignancy within 5 years of randomization, except adequately treated basal cell or squamous cell carcinoma of the skin
* History of a clinically significant reaction to an oligonucleotide compound
* Significant blood loss or blood donation within the 28 days prior to randomization or plasma donation within 7 days prior to randomization
* A tattoo or scarring on the abdomen or any other condition large enough to interfere with the ability to assess injection site reactions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Changes in primary biomarker levels from baseline | Baseline to Day 44
  Changes in polycystin-1 (PC-1) and polycystin-2 (PC-2) protein levels in urinary exosomes from baseline to Day 44

SECONDARY OUTCOMES:
Changes in secondary biomarker levels from baseline | Baseline to Day 44
  Changes in neutrophil gelatinase-associated lipocalin (NGAL) and kidney injury molecule 1 (KIM-1) in urine from baseline to Day 44
Pharmacokinetics (Cmax) | Baseline to Day 44
  Maximum concentration (Cmax) of RGLS4326 in plasma following RGLS4326 treatment
Pharmacokinetics (Tmax) | Baseline to Day 71
  Time to maximum concentration (Tmax) of RGLS4326 in plasma following RGLS4326 treatment
Pharmacokinetics (AUC) | Baseline to Day 71
  Area under the curve (AUC) of RGLS4326 in plasma following RGLS4326 treatment
Number of participants with anti-drug antibodies (ADAs) | Baseline to Day 71
  Incidence of ADAs following RGLS4326 treatment from baseline to Day 71
Titre of anti-drug antibodies (ADAs) in patients with ADAs | Baseline to Day 71
  Titre of ADAs following RGLS4326 treatment from baseline to Day 71
Safety profile | Baseline to Day 71
  Incidence of AEs, lab abnormalities, and ECG abnormalities following RGLS4326 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karl Cremer, PharmD, Study Director — Regulus Therapeutics
Locations (12):
- United States (12):
  - Balboa Nephrology Medical Group, La Mesa, California
  - Academic Medical Research Institute, Los Angeles, California
  - Yale Nephrology Clinical Research, New Haven, Connecticut
  - Accel Research Sites- Mid-Florida Kidney and Hypertension Care, Altamonte Springs, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. Clair Nephrology Research, Roseville, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - UT Southwestern Medical Center, Dallas, Texas
  - ICON Early Phase Services, San Antonio, Texas
  - Swedish Polycystic Kidney Disease Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No